CLINICAL TRIAL: NCT01618578
Title: Comparable Induction of the Rubber Hand Illusion (RHI) in Complex Regional Pain Syndrome Type 1 (CRPS 1) and Healthy Subjects
Brief Title: The Rubber Hand Illusion (RHI) in Patients With CRPS
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof. Dr. med. (Head of the pain clinic of the Bergmannsheil University Hospital), Ruhr University of Bochum
Other Study IDs: RHI2010
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: CRPS; Unilateral Limb Pain of Origin Other Than CRPS
Keywords: rubber hand illusion; CRPS; body image; body ownership

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with CRPS: 24 patients with CRPS of the upper limb type 1 were included into the study.
  Interventions: Procedure: rubber hand illusion
- Patients with unilateral upper limb pain: 21 patients with unilateral upper limb pain served as controls.
  Interventions: Procedure: rubber hand illusion
- healthy subjects: 24 healthy subjects were age- and sex matched to patients with CRPS.
  Interventions: Procedure: rubber hand illusion

INTERVENTIONS:
Procedure: rubber hand illusion — There were three consecutive trials of the RHI:
  1. one control trial: asynchronous condition (3 Min.)
  2. two experimental trials (conducted on both hands):synchronous condition (3 Min.),additionally watching the prosthesis being threatened (20 sec.)

SUMMARY:
The present study investigates by means of the rubber hand illusion body image stability and sense of body ownership in patients with CRPS of the upper limb compared to patients with unilateral pain of origin other than CRPS and age and sex-matched healthy subjects.

DETAILED DESCRIPTION:
In patients with CRPS of the upper limb distortions of body representation and impairments of sense of body ownership are well-known. To investigate the body schema and body image stability of these patients in comparison to patients with upper limb pain of origin other than CRPS and healthy subjects, we conducted a series of rubber hand illusions. This well - established paradigm is elicited by visuo-tactile stimulation of one´s own real hand and a visible hand and forearm prosthesis. The present study investigates 1) if and how far patients with CRPS are susceptible to experience the illusion 2) how far the illusion strength differs between CRPS and patients with unilateral pain of the upper limb of other origin and healthy subjects 3) how far parameters, e.g. neglect-like severity symptoms, body plasticity, empathy, duration of disease and pain intensity influence the illusion strength.

ELIGIBILITY:
Inclusion Criteria:

every participant:

* aged > 18 years
* written informed consent
* free to withdraw participation at any time
* adequate understanding of the german language

Patients with CRPS:

* patients with CRPS type 1 of the upper limb
* clinical symptoms were diagnosed on the basis of the recently modified diagnostic research criteria (Harden, Bruehl et al., 2007)
* proved by typical enhancement in the late phase of the 99m-technetium-triple-phase bone skeleton scintigraphy (Wüppenhorst, Maier et al., 2010)

Patients with unilateral pain of the upper limb:

* unilateral pain
* pain of origin other than CRPS

Healthy subjects:

* age and sex matched to patients with CRPS
* checked by the DFNS IMI questionnaire

Exclusion Criteria:

every participant:

* inadequate understanding of the german language
* missing informed consent
* diabetes mellitus

Patients with CRPS:

-CRPS Type 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study sample consists of three groups:
  1. Patients with CRPS of the upper limb type 1 ( n=24)
  2. Patients with unilateral pain of the upper limb origin other than CRPS (n=21)
  3. Healthy subjects, age and sex-matched to patients with CRPS Patients with unilateral pain of the upper limb of origin other than CRPS serve as controls. Recruitment for all CRPS and the majority of patients in the control group took place in the pain clinic of the Bergmannsheil University Hospital in Bochum. The remaining patients were recruited from the Neurological respectively Surgical department of the Bergmannsheil University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
subjective illusion strength by a validated questionnaire | 1 hour
  The illusion strength was measured subjectively by a validated questionnaire on a 7- point Likert scale,ranging from 0 (= disagree strongly) to 7 (= agree strongly). The questionnaire encompassed five slightly modified items of the German-translated questionnaire by Ocklenburg et al.(2011), following Botvinick & Cohen (1998).In the experimental conditions the questionnaire was additionally augmented by three further statements regarding the perception of the needle threat.

SECONDARY OUTCOMES:
objectified illusion strength by measure of skin conductance response (SCR) | 1 hour
  The SCR represents an objective measure of participant´s identification with the artificial limb, indicating the autonomic nervous system arousal in anticipation of pain, while watching the prosthesis being harmed (Armel & Ramachandran, 2003; Ehrsson, Wiech, Weiskopf, Dolan & Passingham, 2007). In every trial, the SCR was recorded with Ag-AgCl electrodes from the thenar and hypothenar eminence of the non-tested hand. Conductivity was measured in micro-Siemens (1/Ohm).
Measurement of influences of the illusion strength | half an hour
  Several questionnaires were used to assess current and average pain intensity (NRS 0-10), neglect-like severity symptoms (Frettloeh et al. 2006), Handedness (Oldfield,1971), body plasticity (TABP) (Desmond, Horgan et al., 2001), empathy (IRI) ( Davis, 1980) and DASH-score (German, Wind et al. 1999).

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, Prof. Dr., Study Director — Head of the pain clinic of the Bergmannsheil University Hospital
Locations (1):
- Pain clinic of the Bergmannsheil University Hospital, Bochum, Germany